CLINICAL TRIAL: NCT02685124
Title: Metabolomic Approach to Evaluate the Effect of Orange Juice Intake in Healthy Humans: a Comparative Study Between "Bahia" and "Cara Cara" Orange Varieties.
Brief Title: Metabolomic Approach to Evaluate the Effect of Orange Juice Intake in Healthy Humans (METABORANGE).
Acronym: METABORANGE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elisa Brasili, Post doc researcher, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CEP FCF 1097907
Record Dates: First submitted 2016-02-04; First posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bahia orange juice (Experimental): 250 ml twice daily for 7 days
  Interventions: Dietary Supplement: Orange juice
- Cara Cara orange juice (Experimental): 250 ml twice daily for 7 days
  Interventions: Dietary Supplement: Orange juice
- Isocaloric control drink (Placebo Comparator): 250 ml twice daily for 7 days
  Interventions: Dietary Supplement: Orange juice

INTERVENTIONS:
Dietary Supplement: Orange juice — Three days before the start of the study, all participants will restrict their diet avoiding citrus fruits (orange, tangerine, lemon) and its derivatives (washout period), red fruits and vegetables (strawberry, red lettuce, red grape, tomate). The day before the sample collection will be provided a controlled dinner. A fasting for 8 hours will be required before blood and urine collection. All participants will divided into three groups: I (Cara Cara), II (Bahia), III (Isocaloric control drink). They will consume 250 ml of each drink twice daily for 7 consecutive days, with a washout period of 7 days among each intervention.

SUMMARY:
This study evaluates the effect of intake of two orange juice varieties in healthy adults. The participants will receive "Bahia" orange juice, "Cara-Cara" orange juice or a isocaloric control drink in a cross-over study.

DETAILED DESCRIPTION:
The consumption of fruits and vegetables is linked to a decrease in the incidence of chronic diseases. Citrus fruits represent the main source of bioactive compounds such as flavonoids, vitamin C and carotenoids in the brazilian diet.

Unlike the "Bahia", the "Cara Cara" variety which is a spontaneous mutation of "Washington navel" orange is characterized by a bright red pulp due to high levels of lycopene. This difference in the chemical composition may lead to a different biological activity and then a greater protective effect on health.

Since the biological effects generated from a food intake are the result of the interaction of various nutrients with different metabolic pathways, the investigators will apply the metabolomic approach to investigate the complex relationships between fruit intake, bioactive compounds and human metabolism. The investigators will propose to describe the metabolic pathways affected by orange juice intake and to identify biomarkers that can be used in nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects like to drink orange juice

Exclusion Criteria:

* History of cardiovascular disease
* History of gastrointestinal, liver or kidney disease
* History of alcoholism
* Diabetes and metabolic diseases
* Pregnant, trying to became pregnant or breast feeding
* Smokers
* To make use of vitamin and mineral supplements, antibiotics, antiacids, any drugs

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Qualitative changes in urinary metabolome will be evaluated by Gas Chromatography coupled to Mass Spectrometry (GC-MS) and Liquid Chromatography coupled to Mass Spectrometry (LC-MS). | Urine collection will be performed at time 0, after 3, 6 hours and 7 days of treatment.

SECONDARY OUTCOMES:
Changes in the antioxidant enzymes will be evaluated in serum samples in different time points. | Blood collection will be performed at time 0, after 3, 6 hours and 7 days of treatment
Changes in the miRNAs expression will be evaluated in plasma samples in different time points. | Blood collection will be performed at time 0, after 3, 6 hours and 7 days of treatment
Qualitative and quantitative changes in fecal metabolome will be evaluated by an untargeted metabolomic approach based on Nuclear Magnetic Resonance spectroscopy (NMR). | Feces collection will be performed at time 0 and after 7 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Brasili, PhD, Study Director — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: Yes
February 2017